CLINICAL TRIAL: NCT07086027
Title: Clinical, Biochemical, and Microbiological Evaluation of Dental and Periodontal Health in Obese Adolescents: A Cross-Sectional Study
Brief Title: Dental and Periodontal Health in Obese Adolescents: Clinical, Biochemical, and Microbiological Evaluation
Acronym: PERIOBESITY
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-107; Ethics Committee (Other: Marmara University Faculty of Dentistry)
Record Dates: First submitted 2025-07-07; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Obesity; Periodontal Disease; Inflammation Biomarkers; Dental Plaque; Dental Caries
MeSH Terms: conditions — Pediatric Obesity; Periodontal Diseases; Dental Plaque; Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva, serum, GCF, and subgingival plaque samples were collected. DNA was extracted from plaque samples for microbial analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese Group: Adolescents aged 8-13 years with a body mass index (BMI) above the 95th percentile for age and sex, classified as obese. Participants underwent dental examination and provided saliva, serum, gingival crevicular fluid (GCF), and subgingival plaque samples for biomarker and microbiological analysis.
- Control Group (Normal Weight): Adolescents aged 8-13 years with a BMI between the 5th and 85th percentiles for age and sex, considered to have normal weight. The same clinical and sample collection procedures were applied as in the obese group.

SUMMARY:
This study aims to investigate whether obesity affects oral and gum health in children and adolescents. A total of 75 children aged 8 to 13 years participated, including both obese and non-obese individuals. All participants received a dental examination, and samples of saliva, blood, and gum fluid were collected to measure specific inflammation-related substances (such as IL-1α, IL-1β, and leptin). The presence of specific bacteria in the mouth was also analyzed.

DETAILED DESCRIPTION:
This cross-sectional observational study aimed to investigate the relationship between pediatric obesity and periodontal health by integrating clinical, biochemical, and microbiological assessments. A total of 75 adolescents (36 obese and 39 non-obese), aged 8-13 years, were enrolled. Clinical oral evaluations included dft, DMFT, plaque index (PI), gingival index (GI), and probing depth (PD). Blood, saliva, and gingival crevicular fluid (GCF) samples were collected for ELISA-based measurement of pro-inflammatory biomarkers (IL-1α, IL-1β, and leptin). Subgingival plaque samples were analyzed using real-time PCR to quantify six key periodontal pathogens.

ELIGIBILITY:
Inclusion Criteria:

Children aged between 8 and 13 years

Parental consent obtained

No systemic diseases other than obesity

No current medication use

Exclusion Criteria:

Use of antibiotics or anti-inflammatory drugs in the past 3 months

History of systemic disease (other than obesity for the obese group)

Undergoing orthodontic treatment

Missing permanent first molars

Uncooperative behavior during examination

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 75 adolescents aged 8 to 13 years were included in the study. Participants were divided into two groups: obese (BMI > 95th percentile) and normal-weight (BMI 5th-85th percentile). Both groups were evaluated for periodontal status, inflammatory biomarkers, and subgingival microbiota.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Salivary IL-1α Levels | At baseline (single time point, during sample collection visit)
  This outcome measures the concentration of interleukin-1 alpha (IL-1α) in unstimulated saliva and compares levels between obese and non-obese adolescents. Unit of Measure: pg/mL
Salivary IL-1β Levels | At baseline
  This outcome measures the concentration of interleukin-1 beta (IL-1β) in unstimulated saliva and compares levels between obese and non-obese adolescents. Unit of Measure: pg/mL
Salivary Leptin Levels | At baseline
  This outcome measures the concentration of leptin in unstimulated saliva and compares levels between obese and non-obese adolescents. Unit of Measure: pg/mL
Serum IL-1α Levels | At baseline
  This outcome measures the concentration of interleukin-1 alpha (IL-1α) in serum samples and compares levels between obese and non-obese adolescents. Unit of Measure: pg/mL
Serum IL-1β Levels | At baseline
  This outcome measures the concentration of interleukin-1 beta (IL-1β) in serum samples and compares levels between obese and non-obese adolescents. Unit of Measure: pg/mL
Serum Leptin Levels | At baseline
  This outcome measures the concentration of leptin in serum samples and compares levels between obese and non-obese adolescents. Unit of Measure: pg/mL
Gingival Crevicular Fluid (GCF) IL-1α Levels | At baseline
  This outcome measures the concentration of interleukin-1 alpha (IL-1α) in GCF samples and compares levels between obese and non-obese adolescents. Unit of Measure: pg/mL
GCF IL-1β Levels | At baseline
  This outcome measures the concentration of interleukin-1 beta (IL-1β) in GCF samples and compares levels between obese and non-obese adolescents. Unit of Measure: pg/mL
GCF Leptin Levels | At baseline
  This outcome measures the concentration of leptin in GCF samples and compares levels between obese and non-obese adolescents. Unit of Measure: pg/mL
Body Mass Index (BMI) | at baseline
  Unit of Measure: kg/m²
  Description:
  BMI is calculated by dividing weight in kilograms by height in meters squared (kg/m²). Measurements will be used to classify participants as obese (BMI ≥ 95th percentile) or non-obese (BMI < 75th percentile) according to age- and sex-specific CDC growth charts. Higher BMI values indicate greater obesity severity.

SECONDARY OUTCOMES:
Presence of Porphyromonas gingivalis in Subgingival Plaque | At baseline (single time point)
  Detection of P. gingivalis in subgingival plaque samples using real-time PCR. Results will be compared between obese and non-obese adolescents. Unit of Measure: Presence/Absence (or Log genome equivalents if quantitative PCR used)
Presence of Treponema denticola in Subgingival Plaque | At baseline (during clinical examination)
  Detection of reponema denticola in subgingival plaque samples using real-time PCR. Results will be compared between obese and non-obese adolescents. Unit of Measure: Presence/Absence (or Log genome equivalents if quantitative PCR used)
Presence of Tannerella forsythia in Subgingival Plaque | At baseline (during clinical examination)
  Detection of Tannerella forsythia in subgingival plaque samples using real-time PCR. Results will be compared between obese and non-obese adolescents. Unit of Measure: Presence/Absence (or Log genome equivalents if quantitative PCR used)
Presence of Actinobacillus actinomycetemcomitans in Subgingival Plaque | At baseline
  Unit of Measure: Presence/absence (qualitative PCR)
  Description:
  Detection of A. actinomycetemcomitans in subgingival plaque samples using real-time PCR. Results will be compared between obese and non-obese adolescents.
Presence of Prevotella intermedia in Subgingival Plaque | At baseline
  Unit of Measure: Presence/absence (qualitative PCR)
  Description:
  PCR-based detection of P. intermedia in subgingival plaque. Prevalence will be compared between obese and non-obese adolescents.
Presence of Candida albicans in Subgingival Plaque | At baseline
  Unit of Measure: Presence/absence (qualitative PCR)
  Description:
  Identification of Candida albicans in subgingival plaque using real-time PCR and comparison of presence between obese and non-obese groups.
Total Bacterial DNA in Subgingival Plaque | At baseline
  Unit of Measure: Log genome equivalents/sample (quantitative PCR)
  Description:
  Total bacterial DNA load in subgingival plaque will be quantified using real-time PCR and compared between obese and non-obese adolescents.
Plaque Index (PI) Score | At baseline (during clinical examination)
  Unit of Measure: Index score (0-3 scale)
  Description:
  Plaque accumulation will be assessed using the Silness and Löe Plaque Index. Scores range from 0 (no plaque) to 3 (abundant plaque). Higher scores indicate worse oral hygiene.
Gingival Index (GI) Score | At baseline
  Unit of Measure: Index score (0-3 scale)
  Description:
  Gingival inflammation will be evaluated using the Löe and Silness Gingival Index. Scores range from 0 (healthy) to 3 (severe inflammation). Higher scores indicate worse gingival health.
Probing Depth (PD) | At baseline
  Unit of Measure: Millimeters (mm)
  Description:
  Probing depth will be measured at six sites per tooth using a Williams probe. Higher values indicate deeper periodontal pockets and worse periodontal condition.
Bleeding on Probing (BOP) | at baseline
  Unit of Measure: Percentage of sites with bleeding (%)
  Description:
  The proportion of periodontal sites that bleed upon gentle probing will be recorded. Higher percentages indicate greater gingival inflammation.
Dental Caries Experience (dft Index) | At baseline
  Unit of Measure: Number of affected teeth (dft score: 0 to 20)
  Description:
  The dft index (decayed and filled primary teeth) will be recorded to assess caries experience in the primary dentition. Scores range from 0 (no caries experience) to 20 (maximum caries experience in all primary teeth). Higher scores indicate worse dental health.

CONTACTS AND LOCATIONS:
Overall Officials: Çağla Kondoz Torun, DDS, Principal Investigator — Marmara University Faculty of Dentistry Department of Pediatric Dentistry
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) due to ethical and privacy considerations. The study was not designed with data sharing provisions, and participant consent for future data sharing was not obtained.